CLINICAL TRIAL: NCT00815542
Title: Induction of Labor in Oligohydramnios - A Comparison Between Two Modes of Cervical Ripening for Patients With Oligohydramnios at Term
Brief Title: Induction of Labor in Oligohydramnios
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 034-2011-MMC
Record Dates: First submitted 2008-12-25; First posted 2008-12-30 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2012-03

CONDITIONS: Cervical Ripening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- double balloon catheter (Active Comparator): Cervical ripening by double balloon catheter
  Interventions: Device: double balloon catheter
- prostaglandins E2 (Placebo Comparator): cervical ripening using prostaglandins E2
  Interventions: Drug: prostaglandins E2

INTERVENTIONS:
Device: double balloon catheter — cervical ripening using double balloon catheter
  Arms: double balloon catheter
Drug: prostaglandins E2 — prostaglandins E2 - Intravaginal Propess for 24 hours
  Arms: prostaglandins E2

SUMMARY:
When oligohydramnion - decreased amniotic fluid, is diagnosed at term pregnancies, the common practice is to induce labor. Whenever the cervix is not ripened, there are several methods to ripen the cervix, two of which are: mechanical, using a double balloon catheter and pharmacological, with prostaglandins. The aim of the study is to compare those two methods of cervical ripening for patients with significant oligohydramnion at term.

The study will be a prospective randomised trial.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy
* normal pregnancy, well dated, at term
* un ripened cervix

Exclusion Criteria:

* previous cesarean section
* multiple pregnancy
* intra uterine growth restricted fetus

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-06; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Time from ripening to active labor and to delivery, rates of cesarean section, rates of nonreassuring fetal heart rate during induction of labor. | during induction of labor, delivery and early post partum

SECONDARY OUTCOMES:
patients satisfaction | induction of labor, delivery and early postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Tal Biron - Shental, MD, Principal Investigator — Meir Medical Center, Kfar Saba, Israel, Affiliated to Tel Aviv University
Locations (1):
- Meir Medial Center, Kfar Saba, Israel